CLINICAL TRIAL: NCT07089420
Title: ALPCO/Calprotectin CLIA Assay: Expected Values of Calprotectin in Healthy Subjects
Status: Recruiting | Type: Observational
Sponsor: American Laboratory Products Company (Industry)
Responsible Party: Sponsor
Other Study IDs: CPSP-2025-011
Record Dates: First submitted 2025-07-21; First posted 2025-07-28 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: IBD (Inflammatory Bowel Disease); IBS - Irritable Bowel Syndrome; Crohn Disease (CD); UC - Ulcerative Colitis
Keywords: Calprotectin; IBD; IBS
MeSH Terms: conditions — Inflammatory Bowel Diseases; Irritable Bowel Syndrome; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Healthy Adult Volunteers: This group will include approximately 120 to 150 asymptomatic, healthy adults aged 22 years or older. Participants must have no history of inflammatory bowel disease (IBD), irritable bowel syndrome (IBS), gastrointestinal cancer, or chronic intestinal disorders. They must not be taking immunosuppressive therapy, proton pump inhibitors, H2 blockers, or NSAIDs as outlined in the exclusion criteria.
  Participants will collect a single stool sample at home using a provided kit and ship it to the sponsor site (ALPCO) for laboratory analysis. The stool samples will be tested using the ALPCO Calprotectin CLIA assay, a chemiluminescent immunoassay designed to measure fecal calprotectin levels. This group serves to establish reference (expected) calprotectin values in healthy individuals, which will support assay validation and performance claims.
  Interventions: Device: ALPCO Calprotectin CLIA

INTERVENTIONS:
Device: ALPCO Calprotectin CLIA — Measurement of calprotectin in feces

SUMMARY:
This study is evaluating the levels of calprotectin, a protein found in stool, in healthy adults. Calprotectin is a marker of inflammation in the intestines and can help doctors tell the difference between inflammatory bowel diseases (IBD), like Crohn's disease or ulcerative colitis, and non-inflammatory conditions like irritable bowel syndrome (IBS).

In this study, healthy volunteers aged 22 and older will collect a stool sample at home using a simple kit and mail it to the study site. The samples will be tested using a new laboratory method called the ALPCO Calprotectin CLIA assay. The goal is to confirm what level of calprotectin is considered "normal" in people without intestinal disease.

Participation involves just one stool sample, and there are no medical procedures. Volunteers will be compensated for their time. The study will help improve how doctors interpret calprotectin test results in clinical settings.

DETAILED DESCRIPTION:
This study is designed to evaluate the expected (normal) values of calprotectin in the stool of healthy adults using the ALPCO Calprotectin CLIA assay, an investigational in vitro diagnostic test. Calprotectin is a protein released during intestinal inflammation and is commonly used as a non-invasive biomarker to assess gastrointestinal diseases. Elevated levels of fecal calprotectin can indicate active inflammation, particularly in patients with inflammatory bowel disease (IBD), such as Crohn's disease or ulcerative colitis. Conversely, low levels are typically associated with non-inflammatory conditions like irritable bowel syndrome (IBS).

The purpose of this study is to establish baseline (expected) calprotectin levels in individuals who do not have symptoms of IBD, IBS, or other chronic intestinal conditions. These expected values are essential to validate the performance of the ALPCO Calprotectin CLIA assay and to guide its use in differentiating inflammatory and non-inflammatory gastrointestinal conditions in clinical practice.

Approximately 120-150 healthy adult volunteers, aged 22 and older, will be enrolled at 1-2 U.S. clinical sites. Eligible participants will not have any history of chronic intestinal disorders, cancer, recent use of NSAIDs or GI medications, or active gastrointestinal symptoms. After providing informed consent, each participant will collect a stool sample at home using a provided sample collection kit. The sample will be returned to ALPCO by mail or delivery, where it will be analyzed in a laboratory using the study assay.

Stool samples will be processed, stored, and tested according to standardized procedures. The results of this study will be used to determine the reference cut-off value for a healthy population (currently hypothesized at 50 µg/g) and to support the performance claims of the ALPCO Calprotectin CLIA assay in future regulatory submissions.

Participants will be compensated for their participation. There is no direct medical benefit to participants, and the test results will not be shared with them. All samples and data will be handled confidentially, in accordance with Good Clinical Practice (GCP), U.S. FDA regulations, and HIPAA.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥22 years

No abdominal symptoms and no history of inflammatory bowel disease (IBD), irritable bowel syndrome (IBS), or other chronic intestinal disorders

May have undergone colonoscopy with negative findings within the past month or never undergone colonoscopy

Able and willing to provide a stool sample according to the collection protocol

Able to understand the study and sign the informed consent form (ICF)

Exclusion Criteria:

* Unable or unwilling to provide a stool sample

Known active intestinal cancer or history of intestinal cancer with abnormal clinical findings

Currently receiving chemotherapy or systemic immunosuppressive medications

Use of proton pump inhibitors (PPIs) or H2-receptor antagonists within the last 2 weeks

Use of NSAIDs (including aspirin) for 7 or more days in the past 2 weeks

Presence of gastrointestinal symptoms such as abdominal pain, diarrhea, altered appetite, weight loss, or anemia

Samples collected not following protocol requirements

Any other condition that, in the opinion of the investigator, may interfere with study participation or data validity

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will enroll approximately 120 to 150 healthy adult volunteers, aged 22 years or older, from the general U.S. population. Participants must be asymptomatic with no history of inflammatory bowel disease (IBD), irritable bowel syndrome (IBS), gastrointestinal cancer, or other chronic intestinal conditions. Subjects must not be on immunosuppressive therapy, PPIs, H2 blockers, or regular NSAID use prior to sample collection. The goal is to represent a normal, healthy population to establish baseline calprotectin levels using the ALPCO Calprotectin CLIA assay.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-07-07 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Establish the Expected Reference Range for Fecal Calprotectin in Healthy Adults | Within 2 months of sample collection
  Determine the distribution and expected (normal) reference range of fecal calprotectin concentrations in healthy adults using the ALPCO Calprotectin CLIA assay. The outcome will confirm whether the predefined clinical cut-off value of <50 µg/g accurately reflects a non-inflammatory baseline in an asymptomatic population.

CONTACTS AND LOCATIONS:
Locations (1):
- ALPCO, Salem, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No